CLINICAL TRIAL: NCT02231684
Title: A Randomised, Single Centre, Two Period, Incomplete Cross Over Trial in Healthy Subjects Investigating the Pharmacokinetics of Subcutaneous Injections With 1 mg/mL, 3 mg/mL, and 10 mg/mL Semaglutide Strengths and the Absolute Bioavailability of Semaglutide
Brief Title: Investigating the Pharmacokinetics of Subcutaneous Injections With 1 mg/mL, 3 mg/mL, and 10 mg/mL Semaglutide Strengths and the Absolute Bioavailability of Semaglutide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-3687; 2013-004566-34 (EudraCT Number); U1111-1149-3980 (Other: WHO)
Record Dates: First submitted 2014-08-29; First posted 2014-09-04 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- s.c. 0.5 mg (1 mg/ml) followed by s.c. 0.5 mg (3 mg/ml) (Experimental)
  Interventions: Drug: semaglutide
- s.c. 0.5 mg (3 mg/ml) followed by s.c. 0.5 mg (1 mg/ml) (Experimental)
  Interventions: Drug: semaglutide
- s.c. 0.5 mg (3 mg/ml) followed by s.c. 0.5 mg (10 mg/ml) (Experimental)
  Interventions: Drug: semaglutide
- s.c. 0.5 mg (10 mg/ml) followed by s.c. 0.5 mg (3 mg/ml) (Experimental)
  Interventions: Drug: semaglutide
- s.c. 0.5 mg (1 mg/ml) followed by s.c. 0.5 mg (10 mg/ml) (Experimental)
  Interventions: Drug: semaglutide
- s.c. 0.5 mg (10 mg/ml) followed by s.c. 0.5 mg (1 mg/ml) (Experimental)
  Interventions: Drug: semaglutide
- i.v. 0.25 mg (1 mg/ml) followed by s.c. 0.5 mg (1 mg/ml) (Experimental)
  Interventions: Drug: semaglutide
- s.c. 0.5 mg (1 mg/ml) followed by i.v. 0.25 mg (1 mg/ml) (Experimental)
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — Semaglutide administered subcutaneously (s.c. under the skin) in two out of three different strengths (1mg/mL, 3mg/mL and 10 mg/mL).
  Arms: s.c. 0.5 mg (1 mg/ml) followed by s.c. 0.5 mg (10 mg/ml); s.c. 0.5 mg (1 mg/ml) followed by s.c. 0.5 mg (3 mg/ml); s.c. 0.5 mg (10 mg/ml) followed by s.c. 0.5 mg (1 mg/ml); s.c. 0.5 mg (10 mg/ml) followed by s.c. 0.5 mg (3 mg/ml); s.c. 0.5 mg (3 mg/ml) followed by s.c. 0.5 mg (1 mg/ml); s.c. 0.5 mg (3 mg/ml) followed by s.c. 0.5 mg (10 mg/ml)
Drug: semaglutide — Semaglutide administered subcutaneously (s.c. under the skin) in two out of three different strengths (1mg/mL, 3mg/mL and 10 mg/mL) or intravenously (i.v.) (1mg/mL).
  Arms: i.v. 0.25 mg (1 mg/ml) followed by s.c. 0.5 mg (1 mg/ml); s.c. 0.5 mg (1 mg/ml) followed by i.v. 0.25 mg (1 mg/ml)

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the pharmacokinetics (the exposure of the trial drug in the body) of subcutaneous injections of three different strengths of semaglutide and the absolute bioavailability of semaglutide.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects (based on assessment of medical history, physical examination and clinical laboratory data at screening, as judged by the investigator)
* Age between 18 and 55 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 20 and 30 kg/m^2 (both inclusive)

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential not using an adequate contraceptive method. Women of child-bearing potential must use an effective method of birth control for the duration of the trial and for 5 weeks following the last dose of semaglutide. Only highly effective methods of birth control are accepted (i.e. one that results in less than 1 % per year failure rate when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine device) or sexual abstinence or vasectomised partner
* Any clinically significant disease history, in the opinion of the investigator, or systemic or organ disease including: cardiac, pulmonary, gastrointestinal, hepatic, neurologic, renal, genitourinary and endocrine, dermatologic or hematologic diseases
* Use of prescription or non-prescription systemic or topical medicinal products (except routine vitamins, acetylsalicylic acid, paracetamol and contraceptives) within 3 weeks (or within 5 half-lives of the medicinal product, whichever is longest) prior to the first dosing of semaglutide
* History of drug/chemical substance abuse within 1 year from screening, or a positive result in the urine drug test
* History of alcohol abuse within 1 year from screening, or a positive result in the alcohol urine test, or consumption of more than 21 units (male)/14 units (female) of alcohol weekly (one unit of alcohol equals about 250 mL of beer or lager, one glass (120 mL) of wine, or 20 mL spirits)
* Smoking or use of any nicotine products (including nicotine patches, gum etc.) in the last 3 months prior to screening or a positive nicotine test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Area under the semaglutide plasma concentration curve | From day 0-day 35/840 hours

SECONDARY OUTCOMES:
Maximum observed semaglutide plasma concentration | From the concentration-time curves 0 - 840 hours following s.c. administration of a single dose 0.5 mg semaglutide at different strengths
Area under the semaglutide plasma concentration-time curve | From the concentration-time curves 0 - 840 hours following i.v. administration of a single dose 0.25 mg semaglutide (1 mg/mL)
Number of treatment emergent adverse events (TEAEs) | From baseline (Visit 2, Day 1) to follow-up (12-14 weeks after Visit 2)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Berlin, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com